CLINICAL TRIAL: NCT04557696
Title: Implementation and Prospective Evaluation of the REFLECT Communication Curriculum for Oncology Based Medical Graduate Students
Brief Title: A Study to Implement and Evaluate REFLECT Communication Curriculum for Oncology Based Medical Graduate Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resident/fellow feedback indicated study factors made it difficult to participate and busy schedules did not accommodate to consent.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tamara Z. Vern-Gross, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-012188
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Medical Trainees in Oncology Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard oncology curriculum for medical trainees in oncology programs.
- Reflective Group (Experimental): Standard oncology curriculum with standardized patient simulation, in addition to the REFLECT Curriculum workshops for medical trainees in oncology programs.
  Interventions: Other: REFLECT Curriculum

INTERVENTIONS:
Other: REFLECT Curriculum — Annual quarterly workshops will consist of guest lecturers, role playing, patient panels, coaching, knowledge assessments, Standardized Patient (SP) simulations and debriefing/feedback sessions.
  Arms: Reflective Group

SUMMARY:
The purpose of this study is to collect data from quarterly workshops (standardized patient simulations, reflective narratives, questionnaires, surveys, standardized patient and peer feedback, and participant critiques) of participants enrolled in oncology-based residencies and fellowships will be collected. The information that is gathered from this study will be used to describe this population that participate in the workshop and see whether or not introduction of a communication curriculum alongside with the training program will improve communication, self-awareness, and interpersonal skills over time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects: Resident or Fellow enrolled in an oncology related training program (Radiation Oncology, Medical Oncology, Palliative Medicine and Hospice Care, Neurooncology).
* Location: Mayo Clinic Arizona.
* Interest: Willingness to participate.

Exclusion Criteria:

* Schedule does not permit to participation.
* Not enrolled in an oncology-based residency or fellowship at Mayo Clinic Arizona.
* Interest: Not willing to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Emotional Intelligence | Baseline, annually through study completion approximately 10 years
  Change in emotional intelligence comparing baseline scores on the ESCI (Emotional and Social Competence Inventory) with scores on annual ESCI reassessments.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Vern-Gross, DO, FAAP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials